CLINICAL TRIAL: NCT00660296
Title: Randomized Controlled Trial Comparing Co2 vs. Air in Colonoscopy in Sedated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University of Vienna, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EK 07-238-VK
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Pain, Satisfaction
Keywords: CO2; pain; colonoscopy; cancer; screening
MeSH Terms: conditions — Pain; Personal Satisfaction; Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Air insufflation in colonoscopy
  Interventions: Other: Air insufflation use in colonoscopy
- 1 (Other): CO2 insufflation in colonoscopy
  Interventions: Other: CO2 use in colonoscopy

INTERVENTIONS:
Other: Air insufflation use in colonoscopy — Air insufflation for colonic distension
  Arms: 2
Other: CO2 use in colonoscopy — Co2 insufflation for colonic distension
  Arms: 1

SUMMARY:
CO2 insufflation instead of air for colonic distension in colonoscopy is considered to reduce pain after and during colonoscopy. There is limited data, that Co2 is similar effective in sedated patients. Furthermore it had not been investigated if patient's compliance for participating in cancer screening could be improved by using Co2.

The aim of the study is to assess postoperative pain and satisfaction after colonoscopy by comparing C02 with air.

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are assigned to an outdoor ambulance for elective colonoscopy in sedation
* Between 18 and 90 years

Exclusion Criteria:

* COPD
* Dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Pain after Colonoscopy measured by 100mm visual analogue scale. | 15 and 30 minutes and 6 h and 12 h after colonoscopy

SECONDARY OUTCOMES:
patients satisfaction (VAS) and its benefit in regard to cancer screening (2 questions) | 30 minutes and 6 hours after colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, MD, Principal Investigator — Medical University of Vienna; Anton Weiser, MD, Principal Investigator — Ärztezentrum Ost, Anton Baumgartnerstrasse 44, 1230 Vienna
Locations (1):
- Dr. Anton Friedrich Weiser, Vienna, Vienna, Austria

REFERENCES:
- [Result] Bretthauer M, Lynge AB, Thiis-Evensen E, Hoff G, Fausa O, Aabakken L. Carbon dioxide insufflation in colonoscopy: safe and effective in sedated patients. Endoscopy. 2005 Aug;37(8):706-9. doi: 10.1055/s-2005-870154. PMID 16032487